CLINICAL TRIAL: NCT04626531
Title: The Effect of Web-Based Education Program on Metabolic Control, Self-Care Activities, Self-Efficacy and Quality of Life in Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: The Effect of Web-Based Education in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAKU
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2; Educational Problems
Keywords: Nursing; Type 2 diabetes; Web based education program; Self efficacy; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After the pre-tests (Self-Care Activities, Self-Efficacy, Quality of Life) , the patients were given web based education and containing information and recommendations on self-management strategies for three months.
  Interventions: Other: Web-Based Education
- Control Group (Experimental): The control group didn't apply any interference during the study. Participants in the control group continued their routine follow-up.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Web-Based Education — Participants in the intervention group had unlimited access to the Web site, free of charge. The Web site was designed to run on personal computers and smartphones.
  Arms: Intervention Group
Other: Control Group — The control group didn't apply any interference during the study. Participants in the control group continued their routine follow-up.
  Arms: Control Group

SUMMARY:
This research was designed as a randomized controlled study to develop a web-based training program and evaluate the program's impact on diabetes management. This research was carried out on 89 patients diagnosed with type 2 diabetes in the Department of Endocrinology and Metabolic Diseases of Akdeniz University. The preparation of the web page and its content has benefited from the latest literature, national and international websites, and expert opinions. Individuals in the survey scope have been stratified random method with as intervention group (n=44) and control group (n=45). Individuals who were taken in the initiative group were informed by web page, SMS, e-mail prepared for a period of three months. Personal information forms Metabolic Control Variable Form, Diabetes Self-Care Activities Questionnaire, Self-Efficacy Scale for Type 2 Diabetic Individuals, Diabetes-Specific Quality of Life Scale and Web Site Analysis and Measurement Inventory were used as the data tools. The informed consent was obtained from the patients and all data were collected by author during face-to-face interviews.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Diagnosed with type 2 diabetes at least six months ago
* Not have communication disabilities
* Used insulin
* Phone and internet connection

Exclusion Criteria:

* Have a physical, cognitive or mental disability to answer questions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Metabolic Control Variable Form | 5 minute
  It is a 9-item information form that questions the participants' clinical measurements including height, weight, body mass index, blood pressure, and laboratory results including blood glucose, HbA1c, cholesterol, triglyceride, and microalbuminuria level.
The Diabetes Self-Care Activities Questionnaire | 5 minute
  The Diabetes Self-Care Activities Questionnaire was developed by Toobert and Glasgow to determine the self-care activities of individuals with diabetes. The Turkish validity and reliability of the questionnaire were conducted by Kav et al. (2010) and the total Cronbach alpha value was found 0.72. The tool contains 11 items, which measure the frequency of performing dia- betes self-care activities over the last seven days including diet, exercise, blood glucose testing, foot care and tobacco use. The scale total score ranges between 0-7. Higher scores indicate more self-care activities.
The Self-Efficacy Scale for Patients with Type 2 Diabetes Mellitus | 5 minute
  The Self-Efficacy Scale for Patients with Type 2 Diabetes Mellitus was developed in 1999 by Van der Bijl et al. The Turkish validity and reliability of the scale were performed by Kara et al. (2006). The total Cronbach alpha value was found to be 0.88. The scale consists of 20 items in 5-point Likert type. Responses to the scale; "Yes, I'm sure" 5 points "No, I'm not sure" are evaluated as 1 point. The scale total score ranges between 20-100. High scores according to scale total scores indicate good self-efficacy.
The Diabetes Quality of Life Scale | 5 minute
  The Diabetes Quality of Life Scale was developed by Jacobson et al to evaluate the quality of life of individuals with diabetes (Jacobson, Groot, & Samson, 1994). The Turkish validity and reliability study of the scale was conducted by Yıldırım et al (2007). The total Cronbach alpha value of the scale was found to be 0.89. The scale total score ranges between 46-230. High scores according to scale total scores indicate good quality of life.

SECONDARY OUTCOMES:
Website Analysis and Measurement Inventory | 5 minute
  The Website Analysis and Measurement Inventory is a scale based on software evaluation for usability and international software standards. WAMMI is used for the evaluation of websites in many areas. The inventory includes the sub-dimensions of attractiveness, controllability, efficiency, helpfulness, learnability, global usability. The scale total score ranges between 0-100. The scores on the WAMMI are given as percentages, higher percentages indicate higher usability.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal Balci, Proof, Study Chair — Akdeniz University Hospital

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Background] Avdal EU, Kizilci S, Demirel N. The effects of web-based diabetes education on diabetes care results: a randomized control study. Comput Inform Nurs. 2011 Feb;29(2):101-6. doi: 10.1097/NCN.0b013e3181fcbdc6. PMID 21099675
- [Result] Murray E, Sweeting M, Dack C, Pal K, Modrow K, Hudda M, Li J, Ross J, Alkhaldi G, Barnard M, Farmer A, Michie S, Yardley L, May C, Parrott S, Stevenson F, Knox M, Patterson D. Web-based self-management support for people with type 2 diabetes (HeLP-Diabetes): randomised controlled trial in English primary care. BMJ Open. 2017 Sep 27;7(9):e016009. doi: 10.1136/bmjopen-2017-016009. PMID 28954789
- [Result] Yu CH, Parsons JA, Mamdani M, Lebovic G, Hall S, Newton D, Shah BR, Bhattacharyya O, Laupacis A, Straus SE. A web-based intervention to support self-management of patients with type 2 diabetes mellitus: effect on self-efficacy, self-care and diabetes distress. BMC Med Inform Decis Mak. 2014 Dec 14;14:117. doi: 10.1186/s12911-014-0117-3. PMID 25495847